CLINICAL TRIAL: NCT06909318
Title: The Effect of Animated Video and Booklet Education on Asthma Control and Medication Compliance in Children With Asthma: A Randomized Controlled Study
Brief Title: Animated Video and Booklet Education for Improving Asthma Control and Medication Compliance in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Esra Nur Kocaaslan Mutlu, Principal Investigator, Dr. Esra Nur Kocaaslan Mutlu, Assistant Professor of Pediatric Nursing, Trakya University, Trakya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: TUTF-SBF-ENK-06
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Asthma Bronchiale
Keywords: pediatric

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 - Animation Video Group (Experimental): Children receive a 7-minute animated video titled "Living with Asthma" designed for ages 7-11, explaining asthma, its symptoms, triggers, and inhaler techniques through engaging characters. The video is watched initially during a clinic visit and then repeatedly at home with parental guidance over a two-month follow-up period. Parents record viewing frequency using the Parent Observation Form.
  Interventions: Behavioral: Asthma Education - Animated Video
- Arm 2 - Booklet Group (Active Comparator): Children receive a 12-page, illustrated asthma education booklet developed in accordance with GINA guidelines. The booklet is designed with child-friendly visuals and simple language. Parents are instructed to review the booklet with their children at least twice per week over two months and record reading activities using the Parent Observation Form.
  Interventions: Behavioral: Booklet Group
- Arm 3- Control Group (No Intervention): Children receive routine care provided by the Pediatric Allergy and Immunology Outpatient Clinic. This includes standard written forms about allergen avoidance and treatment recommendations based on clinical assessments. No additional asthma education is given during the study period.

INTERVENTIONS:
Behavioral: Asthma Education - Animated Video — This intervention consists of a 7-minute and 39-second animated video titled "Living with Asthma," specifically designed for children aged 7 to 11. The video features two characters, Mert and Robo, who explain asthma, its symptoms, triggers, and correct inhaler techniques in a child-friendly manner. The content is based on the latest GINA (2020) and NHLBI (2020) guidelines. The video is first watched in the clinic setting using a tablet device and then shared with parents via WhatsApp, email, or CD for home viewing. Parents are asked to watch the video with their child at least twice per week for two months and record viewing frequency using a structured observation form. This visual and engaging format distinguishes the intervention from conventional text-based education.
  Arms: Arm 1 - Animation Video Group
Behavioral: Booklet Group — This intervention involves the distribution of a 12-page, full-color, illustrated educational booklet titled "Living with Asthma," developed for children aged 7 to 11. The booklet covers topics such as asthma symptoms, triggers, medication use, and device techniques using simple language and visual aids. Its content was developed in line with GINA (2020) and National Heart, Lung, and Blood Institute (2020) recommendations. During the initial clinic visit, children and parents are introduced to the booklet and instructed to review it together at least twice per week over two months. Parents are also asked to log reading sessions using a structured observation form. This printed, interactive material offers a visually supported, age-appropriate alternative to standard asthma education methods.
  Arms: Arm 2 - Booklet Group

SUMMARY:
Asthma is a chronic inflammatory disease that causes wheezing, coughing, and shortness of breath, and it is a significant cause of morbidity and mortality in the pediatric population. The World Health Organization (WHO) estimated that 262 million people were affected by asthma in 2019, with 461,000 asthma-related deaths annually. In Turkey, the prevalence of asthma in children aged 6-12 ranges from 2% to 16%. Inadequate asthma control in children is often associated with poor medication adherence, lack of knowledge, misbeliefs, and ineffective communication with healthcare professionals. Education is therefore a crucial element of successful asthma management.

Recently, the use of digital tools such as animated videos has become increasingly popular in pediatric education due to their engaging and interactive nature. Studies have shown that visual and interactive materials can improve knowledge, satisfaction, and adherence in children with chronic illnesses.

This randomized controlled study aims to evaluate the effect of an educational intervention using an animated video and booklet on asthma control and medication compliance in children aged 7-11 diagnosed with asthma. It is expected that this child-friendly, visually enriched educational approach will enhance asthma management and support medication adherence in children.

DETAILED DESCRIPTION:
Asthma is a chronic inflammatory airway disease that affects millions of children worldwide and significantly impacts their quality of life, school attendance, and overall health. Despite the availability of effective treatments, asthma control remains suboptimal in many pediatric patients, often due to poor adherence, misinformation, and inadequate education. Educational interventions tailored to children's developmental levels are essential for improving disease management and medication compliance.

This study is designed as a randomized controlled trial to evaluate the impact of an educational program using both an animated video and an illustrated booklet developed specifically for children aged 7 to 11 with a diagnosis of asthma. The intervention focuses on key topics such as asthma triggers, correct inhaler use, symptom recognition, and medication adherence strategies.

Participants will be randomly assigned to either an intervention group receiving the animation and booklet-based education or a control group receiving standard care. Asthma control levels and medication adherence will be measured before and after the intervention using validated scales.

The findings of this study are expected to contribute to the development of child-friendly, visual educational tools that can be used by healthcare professionals in routine asthma care to enhance disease understanding, improve symptom control, and foster treatment adherence in pediatric populations.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 7 and 11 years
* Diagnosed with asthma by a pediatric allergy specialist
* Mild or moderate asthma severity according to GINA criteria
* No communication difficulties
* Have not received any asthma-related education outside of routine clinical care during the study period
* No known mental or neurological disabilities
* No serious chronic illness other than asthma (e.g., cardiac, neurological conditions)
* At least one parent owns a smartphone or tablet
* Child and parent volunteer to participate and provide informed consent

Exclusion Criteria:

* Children younger than 7 or older than 11
* Severe persistent asthma according to GINA criteria
* Communication difficulties
* Prior asthma education outside of routine clinical care
* Children with cognitive or neurological impairments
* Children who frequently require emergency care due to asthma exacerbations
* Families without access to communication tools (e.g., no internet, smartphone, or unable to communicate)
* Lack of consent from either the child or parent

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Asthma control score (Childhood Asthma Control Test - C-ACT) | Baseline, 1st month, and 2nd month follow-up
  Asthma control will be assessed using the Childhood Asthma Control Test (C-ACT), a 7-item validated scale for children aged 4-11. Scores range from 0 to 27. A score ≥20 indicates controlled asthma; ≤19 indicates uncontrolled asthma. It will be administered at baseline, 1st month, and 2nd month follow-up.
Medication Adherence (MARS-5) | Baseline, 1st month, and 2nd month follow-up
  Medication adherence will be measured with the MARS-5 (Medication Adherence Report Scale), a 5-item Likert-type questionnaire. Scores range from 5 to 25; higher scores indicate better adherence. The scale will be administered at baseline, 1st month, and 2nd month.

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya University Faculty of Health Sciences, Edirne, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No